CLINICAL TRIAL: NCT03936088
Title: Use of a Self-Guided Mindfulness Mobile Application to Improve Pain Outcomes in Individuals With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: jilliansylvester (U.S. Federal Agency)
Collaborators: Mike O'Callaghan Military Hospital (U.S. Federal Agency); 375th Medical Group, Scott Air Force Base (U.S. Federal Agency); Travis AFB 60th Med Group (Unknown)
Responsible Party: Sponsor-Investigator, jilliansylvester, Principal Investigator, 375th Medical Group, Scott Air Force Base
Organization: 375th Medical Group, Scott Air Force Base (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FWH20190033H
Record Dates: First submitted 2019-04-30; First posted 2019-05-03 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Osteo Arthritis Knee; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention with Mindfulness App (Headspace) (Experimental): Patient education regarding osteoarthritis, its natural history, and common treatments plus the mindfulness (intervention) app.
  Interventions: Device: Intervention -- "Headspace" mindfulness application
- Control with Water App (My Water Balance) (Active Comparator): Patient education regarding osteoarthritis, its natural history, and common treatments plus the My Water Balance (control) app and provided an in-person demonstration on how to use it.
  Interventions: Device: Control -- "My Water Balance" application

INTERVENTIONS:
Device: Intervention -- "Headspace" mindfulness application — Patients will be provided with a pre-paid 12-week subscription to the mindfulness application, and provided an in-person demonstration on how to use it, and the subscription license code will be recorded for the purposes of tracking use after the conclusion of the study. The intervention group will be asked to use the mindfulness app 10 minutes per day/5 days per week. To standardize Pack usage across all participants, users will be asked to complete the Headspace Essentials", "Pain Management", and "Physical Health" Session Packs.
  Arms: Intervention with Mindfulness App (Headspace)
Device: Control -- "My Water Balance" application — My Water Balance calculates an individual's recommended daily water requirements and assists users in tracking their daily fluid intake. The control group will be asked to log their water intake for the duration of the study, with requested use of 5 days per week to create an equal control. This application is free to download and use. There are options for in-app purchases and application upgrades, though users will be advised against doing so. Information logged in the application may be stored on a third party server; however, no application data will be extracted by the study team. Application use will be reported via weekly surveys, alone.
  Arms: Control with Water App (My Water Balance)

SUMMARY:
This study will investigate if mindfulness training via a smartphone mobile app is effective in improving OA-related knee pain.

DETAILED DESCRIPTION:
The investigator's primary aim in this study is to determine if regular use of a mindfulness application improves pain outcomes in adults with knee osteoarthritis. The investigator's secondary aim is to determine if self-reported Healthcare-Related Quality of Life (HRQoL) scores predict response to mindfulness treatment in OA. The investigators hypothesize that the use of an mHealth intervention for mindfulness training may be an effective adjunct treatment of chronic knee osteoarthritis pain; specifically, that regular use of a mindfulness application will result in a statistically significant reduction in pain outcomes and improvement in physical function as determined by the KOOS scoring system. The investigators also hypothesize that those with lower baseline self-reported HRQoL scores are more likely to see a greater improvement in their pain and function with use of a mindfulness application than those with higher baseline scores.

ELIGIBILITY:
**Patients must be able to get care at Nellis, Scott, or Travis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Male and female Active Duty members and DoD beneficiaries ages 18-74 years
* Meet criteria for symptomatic knee osteoarthritis according to the American College of Rheumatology (pain on more than half of the days of the past month during at least one of the following activities: walking, ascending or descending stairs, standing upright, or lying in bed at night)
* Demonstrate radiographic evidence of OA, with Kellgren and Lawrence (KL) Grade ≥1 as determined by Lead Site Investigator at each study location
* Must have access to a smartphone with enough memory to download the app My Water Balance or the Mindfulness app

Exclusion Criteria:

* Intra-articular corticosteroid injection in the 3 months prior to participation in the study.
* Intra-articular hyaluronic acid/PRP injection in the 6 months prior to participation in the study
* Medical condition contraindicating moderate aerobic exercise as determined by their physician
* History of knee surgery in the past 6 months or previous knee arthroplasty
* Inflammatory joint disease.
* Current Practice of Mindfulness
* Non-English-speaking
* Currently pregnant or planning pregnancy over the study period
* Enrollment in other clinical research study during the study period
* Inability to comply with treatment protocol, including participation in the Rx3 Home Exercise Program.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Post-intervention change in Knee injury and Osteoarthritis Outcome (KOOS) pain subscale | 0,12, 26, 52, and 104 weeks
  The KOOS is a validated knee-specific patient-reported outcome survey designed to assess an individual's perception of their knee pain and associated disability. It has 42 items in 5 separately scored subscales; Pain, other Symptoms, ADL function, Sport and Recreation function, and knee-related Quality of Life (QOL). All items are scored 0-4; for each subscale the scores are transformed to a 0-100 scale (0 representing extreme knee problems and 100 representing no knee problems).

SECONDARY OUTCOMES:
Change in KOOS subscale scores | 0,12, 26, 52, and 104 weeks
  The KOOS is a validated knee-specific patient-reported outcome survey designed to assess an individual's perception of their knee pain and associated disability. It has 42 items in 5 separately scored subscales; Pain, other Symptoms, ADL function, Sport and Recreation function, and knee-related Quality of Life (QOL). All items are scored 0-4; for each subscale the scores are transformed to a 0-100 scale (0 representing extreme knee problems and 100 representing no knee problems).
Change in Five Facet Mindfulness Questionnaire (FFMQ) outcomes | 0,12, 26, 52, and 104 weeks
  The FFMQ-15 is designed to provide a quantitative evaluation of mindfulness. It is based on five independently developed mindfulness questionnaires.The questionnaire has 39 items. The five facets are: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience.
Change in Short Form Health Survey (SF-12) self-reported mental and physical health self-assessments | 0,12, 26, 52, and 104 weeks
  The SF-12 is a generic, multipurpose short-form survey with 12 questions selected from the SF-36 Health Survey which, when combined, scored and weighted, results in two scales of mental and physical functioning and overall health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jillian E Sylvester, MD, Principal Investigator — US Air Force
Locations (1):
- 375th Medical Group, Scott Air Force Base, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan on sharing data

REFERENCES:
- [Background] Ball E, Newton S, Kahan BC, Forbes G, Wright N, Cantalapiedra Calvete C, Gibson HAL, Rogozinska E, Rivas C, Taylor SJC, Birch J, Dodds J. Smartphone App Using Mindfulness Meditation for Women With Chronic Pelvic Pain (MEMPHIS): Protocol for a Randomized Feasibility Trial. JMIR Res Protoc. 2018 Jan 15;7(1):e8. doi: 10.2196/resprot.7720. PMID 29335232
- [Background] Ball EF, Nur Shafina Muhammad Sharizan E, Franklin G, Rogozinska E. Does mindfulness meditation improve chronic pain? A systematic review. Curr Opin Obstet Gynecol. 2017 Dec;29(6):359-366. doi: 10.1097/GCO.0000000000000417. PMID 28961631
- [Background] Cherkin DC, Sherman KJ, Balderson BH, Cook AJ, Anderson ML, Hawkes RJ, Hansen KE, Turner JA. Effect of Mindfulness-Based Stress Reduction vs Cognitive Behavioral Therapy or Usual Care on Back Pain and Functional Limitations in Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA. 2016 Mar 22-29;315(12):1240-9. doi: 10.1001/jama.2016.2323. PMID 27002445
- [Background] Chiesa A, Serretti A. A systematic review of neurobiological and clinical features of mindfulness meditations. Psychol Med. 2010 Aug;40(8):1239-52. doi: 10.1017/S0033291709991747. Epub 2009 Nov 27. PMID 19941676
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] Deshpande BR, Katz JN, Solomon DH, Yelin EH, Hunter DJ, Messier SP, Suter LG, Losina E. Number of Persons With Symptomatic Knee Osteoarthritis in the US: Impact of Race and Ethnicity, Age, Sex, and Obesity. Arthritis Care Res (Hoboken). 2016 Dec;68(12):1743-1750. doi: 10.1002/acr.22897. Epub 2016 Nov 3. PMID 27014966
- [Background] Fish J, Brimson J, Lynch S. Mindfulness Interventions Delivered by Technology Without Facilitator Involvement: What Research Exists and What Are the Clinical Outcomes? Mindfulness (N Y). 2016;7(5):1011-1023. doi: 10.1007/s12671-016-0548-2. Epub 2016 Jun 2. PMID 27642370
- [Background] Fox SD, Flynn E, Allen RH. Mindfulness meditation for women with chronic pelvic pain: a pilot study. J Reprod Med. 2011 Mar-Apr;56(3-4):158-62. PMID 21542535
- [Background] Hootman JM, Helmick CG, Barbour KE, Theis KA, Boring MA. Updated Projected Prevalence of Self-Reported Doctor-Diagnosed Arthritis and Arthritis-Attributable Activity Limitation Among US Adults, 2015-2040. Arthritis Rheumatol. 2016 Jul;68(7):1582-7. doi: 10.1002/art.39692. PMID 27015600
- [Background] IHS Markit, The Complexities of Physician Supply and Demand 2017 Update: Projections from 2016 to 2030. Prepared for the Association of American Medical Colleges. Washington, DC: Association of American Medical Colleges. Accessed November 2018.
- [Background] Jafarzadeh SR, Felson DT. Updated Estimates Suggest a Much Higher Prevalence of Arthritis in United States Adults Than Previous Ones. Arthritis Rheumatol. 2018 Feb;70(2):185-192. doi: 10.1002/art.40355. Epub 2018 Jan 3. PMID 29178176
- [Background] Kotlarz H, Gunnarsson CL, Fang H, Rizzo JA. Insurer and out-of-pocket costs of osteoarthritis in the US: evidence from national survey data. Arthritis Rheum. 2009 Dec;60(12):3546-53. doi: 10.1002/art.24984. PMID 19950287
- [Background] la Cour P, Petersen M. Effects of mindfulness meditation on chronic pain: a randomized controlled trial. Pain Med. 2015 Apr;16(4):641-52. doi: 10.1111/pme.12605. Epub 2014 Nov 7. PMID 25376753
- [Background] Lee AC, Harvey WF, Price LL, Morgan LPK, Morgan NL, Wang C. Mindfulness is associated with psychological health and moderates pain in knee osteoarthritis. Osteoarthritis Cartilage. 2017 Jun;25(6):824-831. doi: 10.1016/j.joca.2016.06.017. Epub 2016 Jun 24. PMID 27349461
- [Background] Lee AC, Harvey WF, Price LL, Han X, Driban JB, Wong JB, Chung M, McAlindon TE, Wang C. Mindfulness Is Associated With Treatment Response From Nonpharmacologic Exercise Interventions in Knee Osteoarthritis. Arch Phys Med Rehabil. 2017 Nov;98(11):2265-2273.e1. doi: 10.1016/j.apmr.2017.04.014. Epub 2017 May 12. PMID 28506776
- [Background] McAlindon TE, LaValley MP, Harvey WF, Price LL, Driban JB, Zhang M, Ward RJ. Effect of Intra-articular Triamcinolone vs Saline on Knee Cartilage Volume and Pain in Patients With Knee Osteoarthritis: A Randomized Clinical Trial. JAMA. 2017 May 16;317(19):1967-1975. doi: 10.1001/jama.2017.5283. PMID 28510679
- [Background] Murphy L, Schwartz TA, Helmick CG, Renner JB, Tudor G, Koch G, Dragomir A, Kalsbeek WD, Luta G, Jordan JM. Lifetime risk of symptomatic knee osteoarthritis. Arthritis Rheum. 2008 Sep 15;59(9):1207-13. doi: 10.1002/art.24021. PMID 18759314
- [Background] Nazarinasab M, Motamedfar A, Moqadam AE. Investigating mental health in patients with osteoarthritis and its relationship with some clinical and demographic factors. Reumatologia. 2017;55(4):183-188. doi: 10.5114/reum.2017.69778. Epub 2017 Aug 31. PMID 29056773
- [Background] Nissen SE, Yeomans ND, Solomon DH, Luscher TF, Libby P, Husni ME, Graham DY, Borer JS, Wisniewski LM, Wolski KE, Wang Q, Menon V, Ruschitzka F, Gaffney M, Beckerman B, Berger MF, Bao W, Lincoff AM; PRECISION Trial Investigators. Cardiovascular Safety of Celecoxib, Naproxen, or Ibuprofen for Arthritis. N Engl J Med. 2016 Dec 29;375(26):2519-29. doi: 10.1056/NEJMoa1611593. Epub 2016 Nov 13. PMID 27959716
- [Background] Skou ST, Roos EM, Laursen MB, Rathleff MS, Arendt-Nielsen L, Simonsen O, Rasmussen S. A Randomized, Controlled Trial of Total Knee Replacement. N Engl J Med. 2015 Oct 22;373(17):1597-606. doi: 10.1056/NEJMoa1505467. PMID 26488691
- [Background] Turner JA, Anderson ML, Balderson BH, Cook AJ, Sherman KJ, Cherkin DC. Mindfulness-based stress reduction and cognitive behavioral therapy for chronic low back pain: similar effects on mindfulness, catastrophizing, self-efficacy, and acceptance in a randomized controlled trial. Pain. 2016 Nov;157(11):2434-2444. doi: 10.1097/j.pain.0000000000000635. PMID 27257859
- [Background] Veehof MM, Trompetter HR, Bohlmeijer ET, Schreurs KM. Acceptance- and mindfulness-based interventions for the treatment of chronic pain: a meta-analytic review. Cogn Behav Ther. 2016;45(1):5-31. doi: 10.1080/16506073.2015.1098724. Epub 2016 Jan 28. PMID 26818413
- [Background] Wang SX, Ganguli AX, Bodhani A, Medema JK, Reichmann WM, Macaulay D. Healthcare resource utilization and costs by age and joint location among osteoarthritis patients in a privately insured population. J Med Econ. 2017 Dec;20(12):1299-1306. doi: 10.1080/13696998.2017.1377717. Epub 2017 Sep 26. PMID 28880733
- [Background] Xie F, Kovic B, Jin X, He X, Wang M, Silvestre C. Economic and Humanistic Burden of Osteoarthritis: A Systematic Review of Large Sample Studies. Pharmacoeconomics. 2016 Nov;34(11):1087-1100. doi: 10.1007/s40273-016-0424-x. PMID 27339668
- [Background] Zangi HA, Mowinckel P, Finset A, Eriksson LR, Hoystad TO, Lunde AK, Hagen KB. A mindfulness-based group intervention to reduce psychological distress and fatigue in patients with inflammatory rheumatic joint diseases: a randomised controlled trial. Ann Rheum Dis. 2012 Jun;71(6):911-7. doi: 10.1136/annrheumdis-2011-200351. Epub 2011 Dec 20. PMID 22186709
- [Background] Zautra AJ, Davis MC, Reich JW, Nicassario P, Tennen H, Finan P, Kratz A, Parrish B, Irwin MR. Comparison of cognitive behavioral and mindfulness meditation interventions on adaptation to rheumatoid arthritis for patients with and without history of recurrent depression. J Consult Clin Psychol. 2008 Jun;76(3):408-421. doi: 10.1037/0022-006X.76.3.408. PMID 18540734

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT03936088/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT03936088/ICF_001.pdf